CLINICAL TRIAL: NCT04702061
Title: Comparison of Erector Spina Plane Block and Thoracic Epidural Block in Breast Surgery
Brief Title: Comparison of Erector Spina Plane Block and Thoracic Epidural Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gulay ERDOGAN KAYHAN, Professor, MD, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Esogu Anesthesia
Record Dates: First submitted 2020-12-24; First posted 2021-01-08 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Breast Neoplasms; Pain, Postoperative
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group E (Active Comparator): Patients who receive general anesthesia after erector spina plane block
  Interventions: Other: Erector spina plane block before general anaesthesia
- Group T (Active Comparator): Patients who receive general anesthesia after thoracic epidural block
  Interventions: Other: Thoracic epidural block before general anaesthesia

INTERVENTIONS:
Other: Erector spina plane block before general anaesthesia — After skin infiltration with 2 ml of 2% lidocaine, an 18 G tuohy needle will be directed between the erector spina muscle and the transverse process of the T4 vertebra using the in-plane technique. The location of the needle will be confirmed by hydrodissection with saline after touching the transverse process. After the plan open, 5 ml of 2% lidocaine, 10 ml of 0.5% bupivacaine and 10 ml of saline, including hydrodissection, will be given in a total amount of 25 ml. Then a 20-G epidural catheter will be inserted 3-4 cm and fixed.
  Arms: Group E
Other: Thoracic epidural block before general anaesthesia — After skin infiltration with 2 ml of 2% lidocaine, an 18 G tuohy needle will be entered through the T4-5 interspinous space (median or paramedian approach). After reaching the thoracic epidural area by loss of resistance method, the epidural catheter will be advanced and fixed to remain 3-4 cm in the epidural area. Following the test dose (2 ml of 2% lidocaine), 3 ml of 2% lidocaine, 5 ml of 0.5% bupivacaine and 5 ml of saline will be administered intermittently in a total volume of 15 ml.
  Arms: Group T

SUMMARY:
The aim of this randomised controlled and double-blind study, is to compare the effects of erector spinae plane (ESP) and thoracic epidural (TEA) blocks on peri-operative hemodynamics and analgesia in patients undergoing unilateral mastectomies due to malignancy.

DETAILED DESCRIPTION:
Patients will be randomised into two groups as Group E (those who received general anesthesia after the erector spina plan block) and Group T (those who received general anesthesia after thoracic epidural block).

After the block skin conductivity (galvanic skin response - GSR), body temperature changes, sympathetic and sensory block levels, peri-operative hemodynamic data, postoperative pain scores and analgesic consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologist) physical classification I-III
* Patients undergoing unilateral mastectomies due to malignancy

Exclusion Criteria:

* Active infection at the intervention site
* History of coagulopathy or anticoagulant use (less time has passed before peripheral and central blocks)
* Major cardiac, pulmonary, renal and neurological diseases
* Autonomic neuropathy or use of drugs that affect autonomic function
* Patients with type 1 diabetes or insulin dependent type 2 diabetes over 10 years
* Allergic to local anesthetics;
* Patients who are uncooperative or have psychiatric problems
* Morbidly obese (body mass index > 35 kg/m2)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Sympathetic block level evaluation with skin conductivity | 45 minutes after block administration
  Skin conductivity will be measured by galvanic skin response (GSR)
Sympathetic block level evaluation with skin temperature | 45 minutes after block administration
  Skin temperature of bilateral thorax will be measured
Sympathetic block level evaluation with hot cold test | 45 minutes after block administration
  Hot cold test of bilateral thorax will be measured
Sympathetic block level evaluation by hemodynamic data | 45 minutes after block administration
  Peri-operative heart rate and mean arterial pressure will be recorded
Sensorial block level evaluation | 45 minutes after block administration
  By pin-prick test

SECONDARY OUTCOMES:
intraoperative hemodynamic data | During the operation
  Heart rate and mean arterial pressure
Postoperative pain scores | 24 hours after operation
  Pain score will be measured with visual analog scale (0-no pain; 10-worst pain) during movement and rest.
Rescue analgesics consumption | During the operation and 24 hours after operation
  Amount of remifentanil (microgram)
Rescue analgesics consumption | 24 hours after operation
  Amount of tramadol (milligram)

CONTACTS AND LOCATIONS:
Overall Officials: Gulay ERDOGAN KAYHAN, MD, Principal Investigator — Professor Doctor
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)